CLINICAL TRIAL: NCT01095029
Title: Cerebral Responses During Bilateral/Unilateral Sacral Nerve Stimulation for Idiopathic Faecal Incontinence - Assessed With Positron Emission Tomography Scan (PET-scan)
Brief Title: Cerebral Responses During Bilateral/Unilateral Sacral Nerve Stimulation for Idiopathic Faecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 003
Record Dates: First submitted 2010-03-22; First posted 2010-03-29 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2012-03

CONDITIONS: Regional Cerebral Blood Flow; Fecal Incontinence
Keywords: Positron emission tomography (PET); Idiopathic Faecal Incontinence; Bilateral Sacral Nerve Stimulation; Sacral Nerve Stimulation; Sacral Nervemodulation
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Off/Off (Experimental): Pacemaker status: Bilateral Off for four weeks before first PET scann.
  Interventions: Device: Medtronic InterStim II - 3058
- On/On (Experimental): Pacemaker status: Bilateral On. PET scan one hour after activation and after four weeks continuous stimulation.
  Interventions: Device: Medtronic InterStim II - 3058
- On/Off (Experimental): Pacemaker status: Unilateral On. PET scan one hour after activation and after four weeks continuous stimulation.
  Interventions: Device: Medtronic InterStim II - 3058

INTERVENTIONS:
Device: Medtronic InterStim II - 3058 — Stimulation with optimal pacemaker settings unilateral and bilateral with standard pacemaker settings: Amplitude sensory treshold, frequency 14 Hz and impulsduration 210 μsec.

SUMMARY:
The purpose of this study is to determine whether Sacral Nerve Stimulation (SNS) for idiopathic faecal incontinence affect cortical and deep brain activity in an acute and chronically stimulation model. Furthermore the association between brain activity and unilateral/bilateral SNS will be studied in each patient. Brain activity will be studied by use of positron emission tomography.

DETAILED DESCRIPTION:
Faecal incontinence is a devastating condition affecting daily living and quality of life. A new treatment Sacral Nerve Stimulation (SNS) has over the last decade given new hope to these patients. In Europe SNS is routinely offered to patients not archiving satisfactory continence result with standard non-surgical treatments. SNS is electrical stimulation of the sacral nerve root(s2,3 or 4). Stimulation of this nerve roots results in improved continence. The mechanism of action is at present not well described. Recent studies have shown that the effect of SNS is by means a neuromodulation in the central nervous system, whereas direct stimulation of efferent nerves to the anal sphincter and the pelvic floor has less significance.

The aim of this study is to describe changes in regional cerebral blood flow (RCBF), with positron emission tomography (PET), in patients implanted bilaterally with sacral neuromodulators with the indication idiopathic faecal incontinence.

RCBF in three deferent stimulations settings will be compared. PET will be performed before and one hour after changes in the activity status of the pacemakers. Four weeks prior to the first scan, patients are informed to switch both neurostimulator off. PET will be performed with the pacemaker settings: OFF/OFF (Stimulation status of left/right pacemaker), On/Off and On/On. The order of the On/OFF and On/On period will be random. Unilateral stimulation will be performed with the pacemaker there has the best efficacy, determined prior to study enrolment. The interval between these three pacemaker settings is four weeks. Four weeks prior to each PET scan the patients fill in bowel habit diaries, bowel habit questionnaires and quality of life assessments.

The association between continence and changes in RCBF will be studied. Additional RCBF and quality of life will be compared.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Informed consent
* Idiopathic fecal incontinence or Fecal incontinence due to small sphincter defect(≤60 o)
* Permanent neuromodulator (medtronic InterStim II) bilateral implanted
* Reduction in fecal incontinence episodes of at least 50% between baseline and latest follow up with unilateral stimulation(Bowel diary card)
* Willing and competent to fill out diary cards
* MR-cerebrum before implantatation of neuromodulator
* Right-handed dominant

Exclusion Criteria:

* Colorectal/proctological surgery since IPG-implant
* Pregnancy
* Neurological diseases including spinal cord injury.
* Use of medication with known alternation of gastrointestinal motilitet (thyroid, diabetes, neuroleptica)
* Claustrofobia
* Latex allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Changes in Regional Cerebral Blood Flow with different pacemaker settings | 12 weeks after study enrolment
  RCBF evaluated with positron emission tomography.

SECONDARY OUTCOMES:
Changes in continence and quality of life with different pacemaker activation. | 12 weeks after study enrolment
  Changes in incontinence episodes and quality of life will be correlated to changes in RCBF with different pacemaker activation.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob K Jakobsen, MD., Principal Investigator — Anal Physiology Laboratory, Surgical Research Section 900, Aarhus University Hospital, Denmark
Locations (1):
- Anal Physiology Laboratory, Surgical Research Section 900, Aarhus University Hospital, Aarhus, Aarhus C, Denmark